CLINICAL TRIAL: NCT02388087
Title: The Iliac Arterio-venous Fistula for Treatment of Neurally Mediated Syncope Study
Acronym: SHAM-ROX NMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Principal Investigator, Neil Sulke, Dr, Eastbourne General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHAM-ROX NMS
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Neurally Mediated Syncope
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ROX COUPLER (Active Comparator): Iliac arterio-venous anastamosis created by insertion of ROX coupler device.
  Interventions: Device: ROX COUPLER
- ROUTINE CARE (Sham Comparator): Right heart catheterisation and Routine care of Neurally mediated syncope.
  Interventions: Procedure: Right heart catheterisation and routine care

INTERVENTIONS:
Device: ROX COUPLER — ROX coupler device is inserted to create an Iliacartero-venous anastamosis following right heart catheterisation.
  Arms: ROX COUPLER
Procedure: Right heart catheterisation and routine care — Participants will have right heart catheterisation followed by routine care. Participants will be blinded to ROX coupler insertion.
  Arms: ROUTINE CARE

SUMMARY:
The purpose of the study is to investigate the efficacy of the ROX coupler in treating patients with tilt test proven Neurally mediated syncope.

DETAILED DESCRIPTION:
Neurally mediated syncope (NMS) is a debilitating condition, with no proven therapeutic measures. The ROX coupler is a device used to create an Iliac arterio-venous anastamosis which allows a shunt of 0.8 litres per minute. The haemodynamic changes following creation of an arterio-venous anastomosis at the iliac level leads to an increase in cardiac preload, reversing finding thought to induce NMS.

This a randomised controlled study to evaluate the effect of Iliac arterio-venous anastamosis in patients with neurally mediated syncope. The Head up tilt test is used as an objective measure to evaluate the effect of the arterio-venous anastamosis in patients with NMS. Participants with tilt test proven NMS will be eligible for the study ( if they satisfy all other eligibility criteria). Participants will be randomised to ROX coupler intervention or standard therapy. The primary outcome measure will be absence of loss consciousness on tilt table testing at 3 months post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Absence of transient loss of consciousness associated with reflex bradycardia or hypotension on tilt testing at 3 months following randomised intervention

Exclusion Criteria:

* Time to first episode of syncope after randomised intervention
* Number of syncopal episodes in the first 3 months after randomised intervention.
* Tilt table response at 6 months following randomised intervention i.e. 3 months after unblinding
* Number of syncopal episodes at 6 months after intervention i.e. 3 months after unblinding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Absence of loss of consciousness on tilt table testing | 3 months
  Absence of loss of consciousness associated with reflex bradycardia or hypotension on head up tilt table testing at 3 months post intervention

SECONDARY OUTCOMES:
Time to first episode of syncope after randomised intervention | 3 months
Number of syncopal episodes in the first 3 months after randomised intervention | 3 months
Tilt table response at 6 months following randomised intervention i.e. 3 months after unblinding | 6 months
Number of syncopal episodes at 6 months after intervention i.e. 3 months after unblinding | 6 months

OTHER OUTCOMES:
Heart rate variability following intervention as observed on 24 hour holter monitoring | 3 and 6 months
Changes in echocardiographic parameters following intervention compared to baseline. | 3 and 6months
Change in exercise capacity assessed by cardio-pulmonary exercise testing after intervention compared to baseline. | 3 and 6months